CLINICAL TRIAL: NCT07370220
Title: Rutin Therapy Reduces Ulcerative Colitis Disease Activity By Inhibiting The NOD-Like Receptor Protein 3 (NLRP3) Inflammasome: A Molecular Assessment in an Interventional Study.
Brief Title: Effect of Rutin on Inflammation Pathways in Ulcerative Colitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Raafat R. Mohammed, Assistant consultant of Clinical Pathology, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Rc 3.1.2025
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Rutin; Tablets

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Ulcerative Colitis (UC-A) (Active Comparator)
  Interventions: Drug: Rutin 500 MG Oral Tablet; Diagnostic Test: Fecal Calprotectin
- Remission Ulcerative Colitis (UC-B) (Active Comparator)
  Interventions: Diagnostic Test: Fecal Calprotectin; Drug: Placebo
- Healthy Control (Group C) (Placebo Comparator)
  Interventions: Diagnostic Test: Fecal Calprotectin

INTERVENTIONS:
Drug: Rutin 500 MG Oral Tablet — Oral capsules twice daily for 30 days
  Arms: Active Ulcerative Colitis (UC-A)
Diagnostic Test: Fecal Calprotectin — Sample collection only for baseline comparison.
Drug: Placebo — Placebo tablets for 30 days
  Arms: Remission Ulcerative Colitis (UC-B)

SUMMARY:
This study evaluates the therapeutic role of Rutin (a plant-derived flavonoid) in reducing the severity of Ulcerative Colitis (UC). The study investigates whether Rutin can decrease intestinal inflammation and improve clinical symptoms by inhibiting the NLRP3 inflammasome signaling pathway, which is activated by oxidative stress in the colon.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC confirmed by endoscopy/histology.
* Age 18 to 65 years.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Known hypersensitivity to Rutin.
* Presence of other serious systemic diseases (e.g., malignancy, severe hepatic or renal failure).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-22 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Success Rate of Clinical Improvement | Day 30 (End of treatment)
  The percentage of participants who achieve clinical improvement at the end of the treatment period. Clinical improvement is defined as reaching a score of 5 or less on the Simple Clinical Colitis Activity Index (SCCAI).

SECONDARY OUTCOMES:
Change in Fecal Calprotectin Levels | Baseline and Day 30
  The concentration of Fecal Calprotectin measured in stool samples to quantify the reduction in intestinal inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha Faculty of Medicine, Banhā, Al Qalyoubia, Egypt